CLINICAL TRIAL: NCT02843971
Title: Evaluation of the Water Drinking Test Response in Supine and Sitting Position Using the Continuous Intraocular Pressure Measurement Device Sensimed Triggerfish in Healthy Subjects
Brief Title: Evaluation of the Water Drinking Test Response in Supine and Sitting Position Using the Continuous Measurement Device Sensimed Triggerfish Intraocular Pressure in Healthy Subjects
Acronym: PIO-WDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC14.317
Record Dates: First submitted 2015-01-13; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-06

CONDITIONS: Intraocular Pressure
Keywords: Water Drinking Test; Intraocular Pressure; Sensimed Triggerfish
MeSH Terms: interventions — Tonometry, Ocular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy volunteers (Experimental)
  Interventions: Device: Intraocular pressure measurement with the Sensimed triggerfish Device

INTERVENTIONS:
Device: Intraocular pressure measurement with the Sensimed triggerfish Device

SUMMARY:
Monocentric, prospective study, comparison of the water drinking test response in the supine and in the sitting position using the intraocular pressure monitoring device Sensimed Triggerfish in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Aged over 18 years
* No previous ophthalmic conditions
* Spherical equivalent from - 6 to +3 diopters

Exclusion Criteria:

* Contact lens use

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Measure of intraocular pressure while lying down | 30 minutes
  Peak IOP defined by the maximum level reached Peak period defined by the time from the ingestion of water and the occurrence of the IOP; and Time to get back to the initial pressure, as measured with the sensimed triggerfish device.
  On one eye and the lens is inserted on the other eye.
Measure of intraocular pressure while sitting | 30 minutes
  Peak IOP defined by the maximum level reached; Peak period defined by the time from the ingestion of water and the occurrence of the IOP; and Time to get back to the initial pressure, as measured with the sensimed triggerfish device.
  On one eye and the lens is inserted on the other eye.
Measure of intraocular pressure on the eye without the lens. | 30 minutes
  Peak IOP defined by the maximum level reached; Peak period defined by the time from the ingestion of water and the occurrence of the IOP; and Time to get back to the initial pressure, as measured with the non-contact tonometer.
Mesure of intraocular pressure on the eye | One hour and a half
  Six results. Without the lens each 15 minutes. After drinking 1 L of water.
Mesure of intraocular pressure on the eye without the lens each 30 minutes. | One hour
  Two results. After drinking 1 L of water.

CONTACTS AND LOCATIONS:
Overall Officials: Florent APTEL, MD, PhD, Principal Investigator — Department of Ophthalmology CHU de Grenoble/University Hospital of Grenoble
Locations (1):
- University Hospital of Grenoble, Grenoble, France

REFERENCES:
- [Background] Quigley HA, Broman AT. The number of people with glaucoma worldwide in 2010 and 2020. Br J Ophthalmol. 2006 Mar;90(3):262-7. doi: 10.1136/bjo.2005.081224. PMID 16488940
- [Background] Guo L, Moss SE, Alexander RA, Ali RR, Fitzke FW, Cordeiro MF. Retinal ganglion cell apoptosis in glaucoma is related to intraocular pressure and IOP-induced effects on extracellular matrix. Invest Ophthalmol Vis Sci. 2005 Jan;46(1):175-82. doi: 10.1167/iovs.04-0832. PMID 15623771
- [Background] Fuchshofer R. The pathogenic role of transforming growth factor-beta2 in glaucomatous damage to the optic nerve head. Exp Eye Res. 2011 Aug;93(2):165-9. doi: 10.1016/j.exer.2010.07.014. Epub 2010 Aug 12. PMID 20708611
- [Background] Leske MC, Wu SY, Hennis A, Honkanen R, Nemesure B; BESs Study Group. Risk factors for incident open-angle glaucoma: the Barbados Eye Studies. Ophthalmology. 2008 Jan;115(1):85-93. doi: 10.1016/j.ophtha.2007.03.017. Epub 2007 Jul 16. PMID 17629563
- [Background] Le A, Mukesh BN, McCarty CA, Taylor HR. Risk factors associated with the incidence of open-angle glaucoma: the visual impairment project. Invest Ophthalmol Vis Sci. 2003 Sep;44(9):3783-9. doi: 10.1167/iovs.03-0077. PMID 12939292
- [Background] Gordon MO, Beiser JA, Brandt JD, Heuer DK, Higginbotham EJ, Johnson CA, Keltner JL, Miller JP, Parrish RK 2nd, Wilson MR, Kass MA. The Ocular Hypertension Treatment Study: baseline factors that predict the onset of primary open-angle glaucoma. Arch Ophthalmol. 2002 Jun;120(6):714-20; discussion 829-30. doi: 10.1001/archopht.120.6.714. PMID 12049575
- [Background] European Glaucoma Prevention Study (EGPS) Group; Miglior S, Pfeiffer N, Torri V, Zeyen T, Cunha-Vaz J, Adamsons I. Predictive factors for open-angle glaucoma among patients with ocular hypertension in the European Glaucoma Prevention Study. Ophthalmology. 2007 Jan;114(1):3-9. doi: 10.1016/j.ophtha.2006.05.075. Epub 2006 Oct 27. PMID 17070596
- [Background] Sommer A, Tielsch JM, Katz J, Quigley HA, Gottsch JD, Javitt J, Singh K. Relationship between intraocular pressure and primary open angle glaucoma among white and black Americans. The Baltimore Eye Survey. Arch Ophthalmol. 1991 Aug;109(8):1090-5. doi: 10.1001/archopht.1991.01080080050026. PMID 1867550
- [Background] Kass MA, Heuer DK, Higginbotham EJ, Johnson CA, Keltner JL, Miller JP, Parrish RK 2nd, Wilson MR, Gordon MO. The Ocular Hypertension Treatment Study: a randomized trial determines that topical ocular hypotensive medication delays or prevents the onset of primary open-angle glaucoma. Arch Ophthalmol. 2002 Jun;120(6):701-13; discussion 829-30. doi: 10.1001/archopht.120.6.701. PMID 12049574
- [Background] Miglior S, Zeyen T, Pfeiffer N, Cunha-Vaz J, Torri V, Adamsons I; European Glaucoma Prevention Study (EGPS) Group. Results of the European Glaucoma Prevention Study. Ophthalmology. 2005 Mar;112(3):366-75. doi: 10.1016/j.ophtha.2004.11.030. PMID 15745761
- [Background] The Advanced Glaucoma Intervention Study (AGIS): 7. The relationship between control of intraocular pressure and visual field deterioration.The AGIS Investigators. Am J Ophthalmol. 2000 Oct;130(4):429-40. doi: 10.1016/s0002-9394(00)00538-9. PMID 11024415
- [Background] Heijl A, Leske MC, Bengtsson B, Hyman L, Bengtsson B, Hussein M; Early Manifest Glaucoma Trial Group. Reduction of intraocular pressure and glaucoma progression: results from the Early Manifest Glaucoma Trial. Arch Ophthalmol. 2002 Oct;120(10):1268-79. doi: 10.1001/archopht.120.10.1268. PMID 12365904
- [Background] The effectiveness of intraocular pressure reduction in the treatment of normal-tension glaucoma. Collaborative Normal-Tension Glaucoma Study Group. Am J Ophthalmol. 1998 Oct;126(4):498-505. doi: 10.1016/s0002-9394(98)00272-4. PMID 9780094
- [Background] Mosaed S, Liu JH, Weinreb RN. Correlation between office and peak nocturnal intraocular pressures in healthy subjects and glaucoma patients. Am J Ophthalmol. 2005 Feb;139(2):320-4. doi: 10.1016/j.ajo.2004.09.062. PMID 15733994
- [Background] Liu JH, Kripke DF, Hoffman RE, Twa MD, Loving RT, Rex KM, Gupta N, Weinreb RN. Nocturnal elevation of intraocular pressure in young adults. Invest Ophthalmol Vis Sci. 1998 Dec;39(13):2707-12. PMID 9856781
- [Background] Hara T, Hara T, Tsuru T. Increase of peak intraocular pressure during sleep in reproduced diurnal changes by posture. Arch Ophthalmol. 2006 Feb;124(2):165-8. doi: 10.1001/archopht.124.2.165. PMID 16476884
- [Background] Asrani S, Zeimer R, Wilensky J, Gieser D, Vitale S, Lindenmuth K. Large diurnal fluctuations in intraocular pressure are an independent risk factor in patients with glaucoma. J Glaucoma. 2000 Apr;9(2):134-42. doi: 10.1097/00061198-200004000-00002. PMID 10782622
- [Background] Nouri-Mahdavi K, Hoffman D, Coleman AL, Liu G, Li G, Gaasterland D, Caprioli J; Advanced Glaucoma Intervention Study. Predictive factors for glaucomatous visual field progression in the Advanced Glaucoma Intervention Study. Ophthalmology. 2004 Sep;111(9):1627-35. doi: 10.1016/j.ophtha.2004.02.017. PMID 15350314
- [Background] Caprioli J, Coleman AL. Intraocular pressure fluctuation a risk factor for visual field progression at low intraocular pressures in the advanced glaucoma intervention study. Ophthalmology. 2008 Jul;115(7):1123-1129.e3. doi: 10.1016/j.ophtha.2007.10.031. Epub 2008 Feb 20. PMID 18082889
- [Background] Liu JH, Kripke DF, Twa MD, Hoffman RE, Mansberger SL, Rex KM, Girkin CA, Weinreb RN. Twenty-four-hour pattern of intraocular pressure in the aging population. Invest Ophthalmol Vis Sci. 1999 Nov;40(12):2912-7. PMID 10549652
- [Background] Sit AJ, Weinreb RN, Crowston JG, Kripke DF, Liu JH. Sustained effect of travoprost on diurnal and nocturnal intraocular pressure. Am J Ophthalmol. 2006 Jun;141(6):1131-3. doi: 10.1016/j.ajo.2006.01.049. PMID 16765686
- [Background] Romanet JP, Maurent-Palombi K, Noel C, Bourdon L, Pepin JL, Mouillon M, Buguet A. [Nyctohemeral variations in intraocular pressure]. J Fr Ophtalmol. 2004 Sep;27 Spec No 2:2S19-2S26. French. PMID 15314571
- [Background] Hjortdal JO, Jensen PK. In vitro measurement of corneal strain, thickness, and curvature using digital image processing. Acta Ophthalmol Scand. 1995 Feb;73(1):5-11. doi: 10.1111/j.1600-0420.1995.tb00004.x. PMID 7627759
- [Background] Mansouri K, Shaarawy T. Continuous intraocular pressure monitoring with a wireless ocular telemetry sensor: initial clinical experience in patients with open angle glaucoma. Br J Ophthalmol. 2011 May;95(5):627-9. doi: 10.1136/bjo.2010.192922. Epub 2011 Jan 7. PMID 21216796
- [Background] De Smedt S, Mermoud A, Schnyder C. 24-hour intraocular pressure fluctuation monitoring using an ocular telemetry Sensor: tolerability and functionality in healthy subjects. J Glaucoma. 2012 Oct-Nov;21(8):539-44. doi: 10.1097/IJG.0b013e31821dac43. PMID 21602707
- [Background] Mansouri K, Medeiros FA, Tafreshi A, Weinreb RN. Continuous 24-hour monitoring of intraocular pressure patterns with a contact lens sensor: safety, tolerability, and reproducibility in patients with glaucoma. Arch Ophthalmol. 2012 Dec;130(12):1534-9. doi: 10.1001/jamaophthalmol.2013.1350. PMID 23229696
- [Background] Freiberg FJ, Lindell J, Thederan LA, Leippi S, Shen Y, Klink T. Corneal thickness after overnight wear of an intraocular pressure fluctuation contact lens sensor. Acta Ophthalmol. 2012 Nov;90(7):e534-9. doi: 10.1111/j.1755-3768.2012.02495.x. Epub 2012 Sep 13. PMID 22974389
- [Background] Pajic B, Pajic-Eggspuchler B, Haefliger I. Continuous IOP fluctuation recording in normal tension glaucoma patients. Curr Eye Res. 2011 Dec;36(12):1129-38. doi: 10.3109/02713683.2011.608240. Epub 2011 Oct 6. PMID 21978205
- [Background] Mansouri K, Liu JH, Weinreb RN, Tafreshi A, Medeiros FA. Analysis of continuous 24-hour intraocular pressure patterns in glaucoma. Invest Ophthalmol Vis Sci. 2012 Dec 13;53(13):8050-6. doi: 10.1167/iovs.12-10569. PMID 23139273
- [Background] Lorenz K, Korb C, Herzog N, Vetter JM, Elflein H, Keilani MM, Pfeiffer N. Tolerability of 24-hour intraocular pressure monitoring of a pressure-sensitive contact lens. J Glaucoma. 2013 Apr-May;22(4):311-6. doi: 10.1097/IJG.0b013e318241b874. PMID 23524857
- [Background] Hubanova R, Aptel F, Chiquet C, Mottet B, Romanet JP. Effect of overnight wear of the Triggerfish((R)) sensor on corneal thickness measured by Visante((R)) anterior segment optical coherence tomography. Acta Ophthalmol. 2014 Mar;92(2):e119-23. doi: 10.1111/aos.12241. Epub 2013 Jul 15. PMID 23848265
- [Background] Mottet B, Aptel F, Romanet JP, Hubanova R, Pepin JL, Chiquet C. 24-hour intraocular pressure rhythm in young healthy subjects evaluated with continuous monitoring using a contact lens sensor. JAMA Ophthalmol. 2013 Dec;131(12):1507-16. doi: 10.1001/jamaophthalmol.2013.5297. PMID 24158696
- [Background] Danesh-Meyer HV. The water-drinking test: the elegance of simplicity. Clin Exp Ophthalmol. 2008 May;36(4):301-3. doi: 10.1111/j.1442-9071.2008.01782.x. No abstract available. PMID 18700912
- [Background] Friberg TR, Sanborn G, Weinreb RN. Intraocular and episcleral venous pressure increase during inverted posture. Am J Ophthalmol. 1987 Apr 15;103(4):523-6. doi: 10.1016/s0002-9394(14)74275-8. PMID 3565513
- [Background] Diestelhorst M, Krieglstein GK. The effect of the water-drinking test on aqueous humor dynamics in healthy volunteers. Graefes Arch Clin Exp Ophthalmol. 1994 Mar;232(3):145-7. doi: 10.1007/BF00176783. PMID 8188063
- [Background] Hayreh SS. Acute occlusive disorders of the choroidal vasculature. Int Ophthalmol. 1983 Feb;6(2):139-48. doi: 10.1007/BF00127642. No abstract available. PMID 6682094
- [Background] Kumar RS, de Guzman MH, Ong PY, Goldberg I. Does peak intraocular pressure measured by water drinking test reflect peak circadian levels? A pilot study. Clin Exp Ophthalmol. 2008 May;36(4):312-5. doi: 10.1111/j.1442-9071.2008.01765.x. PMID 18700916
- [Background] MILLER D. THE RELATIONSHIP BETWEEN DIURNAL TENSION VARIATION AND THE WATER-DRINKING TEST. Am J Ophthalmol. 1964 Aug;58:243-6. doi: 10.1016/0002-9394(64)91571-5. No abstract available. PMID 14204331
- [Background] Frankelson EN. The role of the water test in evaluation of glaucoma control. Can J Ophthalmol. 1974 Oct;9(4):408-10. No abstract available. PMID 4473065
- [Background] Chen CH, Lu DW, Chang CJ, Chiang CH, Chou PI. The application of water drinking test on the evaluation of trabeculectomy patency. J Ocul Pharmacol Ther. 2000 Feb;16(1):37-42. doi: 10.1089/jop.2000.16.37. PMID 10673129
- [Background] Hubanova R, Aptel F, Zhou T, Arnol N, Romanet JP, Chiquet C. Comparison of intraocular pressure measurements with the Reichert Pt100, the Keeler Pulsair Intellipuff portable noncontact tonometers, and Goldmann applanation tonometry. J Glaucoma. 2015 Jun-Jul;24(5):356-63. doi: 10.1097/01.ijg.0000435776.99193.41. PMID 24240887
- [Background] Aptel F, Tamisier R, Pepin JL, Mottet B, Hubanova R, Romanet JP, Chiquet C. Hourly awakening vs continuous contact lens sensor measurements of 24-hour intraocular pressure: effect on sleep macrostructure and intraocular pressure rhythm. JAMA Ophthalmol. 2014 Oct;132(10):1232-8. doi: 10.1001/jamaophthalmol.2014.1761. PMID 25074578
- [Background] Susanna R Jr, Hatanaka M, Vessani RM, Pinheiro A, Morita C. Correlation of asymmetric glaucomatous visual field damage and water-drinking test response. Invest Ophthalmol Vis Sci. 2006 Feb;47(2):641-4. doi: 10.1167/iovs.04-0268. PMID 16431962